CLINICAL TRIAL: NCT04916496
Title: Effect of Acceptance and Commitment Therapy-based Lifestyle Counselling Programme for People With Early Psychosis on Physical Activity: A Pilot Randomised Controlled Trial
Brief Title: Acceptance and Commitment Therapy-based Lifestyle Counselling Programme for Early Psychosis on Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: North District Hospital (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05190027
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Acceptance and Commitment Therapy; Randomised Controlled Trial; Lifestyle Counselling Programme; Psychosis; Physical Activity
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; repeated-measures 2-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and researchers(and health care providers of the study hospital) are blinded to the group assignment and intervention undertaken and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-LCP Group (Experimental): An Acceptance and Commitment Therapy-based healthy lifestyle counselling programme (ACT-LCP) and routine psychiatric outpatient/rehabilitation services of the study hospital.
  Interventions: Behavioral: Acceptance and Commitment Therapy-based lifestyle counselling programme
- Control Group (Placebo Comparator): A healthy lifestyle talk and routine psychiatric outpatient/rehabilitation services of the study hospital.
  Interventions: Behavioral: Healthy lifestyle talk

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy-based lifestyle counselling programme — The ACT-LCP Group will receive an ACT-based lifestyle counselling programme, which composes of 5-weekly group sessions (2 hours per each, 15 hours in total). Acceptance, mindfulness, values clarification skills/exercises will be used to help patients to increase self-perspective taking and willingness to experience distressing sensations, discomfort and urges while engaging in healthy lifestyle behaviours.
  One month after the programme, the participant will receive one 'booster' session (2 hours), followed by 2-weekly telephone follow-up calls (20-30 minutes per call) to evaluate the effort of behavioural change.
  Arms: ACT-LCP Group
Behavioral: Healthy lifestyle talk — The Control Group will receive one 2-hour, healthy lifestyle education talk (at least 10 patients in the talk) based on the HEARTS technical package as recommended by the WHO as routine care. This package includes a collection of evidence-based protocols which standardizes a clinical approach to promote a healthy lifestyle among adults. The Control Group will receive routine psychiatric outpatient/rehabilitation services as provided by the clinic in NDH/community centre.
  One month after the talk, three weekly follow-up telephone calls (20-30 minutes) will be arranged for each patient in the Control Group to evaluate the effort of behavioural change.
  Arms: Control Group

SUMMARY:
This pilot randomized controlled trial aims to determine the feasibility, acceptability and preliminary effects of an Acceptance and Commitment Therapy-based Lifestyle Counselling Programme (ACT-LCP) on the physical and psychosocial health outcomes of patients with early psychosis over a 12-week follow-up.

DETAILED DESCRIPTION:
Background: Three-quarters of deaths in psychotic patients are caused by Cardiometabolic Diseases (CMD), including but not limited to cardiac disease, diabetes, and stroke. Globally, the average life expectancy of a psychotic patient is 10 to 20 years shorter than the average life expectancy of those without a psychotic diagnosis. Research has supported that early intervention on lifestyle and cardiometabolic risks is essential to prevent the occurrence of CMD. This study will integrate the framework of Acceptance and Commitment Therapy and Self-Determination Therapy with a healthy-lifestyle intervention programme cultivating autonomous motivation of psychotic patients to live healthier. In addition, the acceptance and mindfulness-based part of ACT would increase the patient's awareness to psychological struggles. While many studies reviewed the ACT's effectiveness in improving mental health and functioning outcomes as well as enhancing physical activity and maintenance of weight reduction for individuals without mental illness, the use of the ACT-based lifestyle intervention in psychotic patients with the framework of Self-Determination Therapy has not even been examined.

Objectives: To determine the feasibility, acceptability and preliminary effects of an Acceptance and Commitment Therapy-based Lifestyle Counselling Programme (ACT-LCP) on the physical and psychosocial health outcomes of patients with early psychosis over a 12-weeks follow-up period.

Hypotheses to be tested: When compared with the Control Group receiving standard care and lifestyle education talk, more participants in the ACT-LCP Group will be physically active, defined as participating in at least 150 minutes/week of moderate to vigorous-intensity of physical activity, at 1-week and at 12-weeks post-intervention. The ACT-LCP group will report improvements in healthy dietary intake, autonomous motivation, psychological flexibility, mental status and quality of life.

Design and subjects: An assessor-blind randomized controlled trial with two-arm, repeated-measures design; 72 Cantonese-speaking patients with early psychosis.

Study Instruments: Validated questionnaires, accelerometer-based wristband activity tracker

Intervention: One ACT-LCP, including 5-weekly sessions (2 hours/session) of group therapy, one 'booster' session to be held at 1-month afterwards, followed by 2-weekly telephone follow-ups.

Main outcome measure: Prevalence of being physically active, as measured by the accelerometer-based wristband activity tracker at 12 weeks post-intervention.

Data analysis: The assessment of acceptability and feasibility of the ACT-LCP will be assessed by examining the recruitment rate, the attrition rate, the completion of after-session homework and post programme focus group interviews. Generalized estimating equations with covariate adjustments will be used to examine the preliminary effects of ACT-LCP.

Expected results: Patients with early psychosis will become more autonomously motivated and more psychologically flexible to continue regular healthy lifestyle behaviours, leading to improvements in health outcomes.

ELIGIBILITY:
Inclusion criteria:

1. at least 18 years of age or above
2. able to understand the nature of the study and give informed consent,
3. able to communicate in Cantonese,
4. have a diagnosis of psychotic disorders (e.g., delusional/brief psychotic disorder, schizotypal disorder, and psychosis not otherwise specified) according to the DSM IV-TR, DSM-V or ICD-10, within 5 years of onset as documented in their clinical/written records;
5. insufficiently active (i.e., <150 minutes of MVPA per week) based on self-reports in a brief screening form, and
6. having used mobile instant-messaging apps (e.g. WhatsApp/Facebook messenger/WeChat) installed on a smartphone.

Exclusion criteria:

1. have had a record of alcohol abuse and/or substance misuse,
2. poor physical health condition, acute/severe medical diseases seriously reducing their life expectancy or ability to participate,
3. pregnancy or within six months of postpartum,
4. have received (within the past 6 months) or are receiving other physical and psychosocial interventions, and
5. severe psychiatric symptoms appeared in the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change from baseline assessment to 12 weeks post-intervention
  An accelerometer-based wristband activity tracker, the Fitbit Inspire 2, will be used to measure the total number of minutes spent on moderate to vigorous physical activity (MVPA). Examples of MVPA include brisk walking, climbing stairs, dancing or doing household chores (moderate activity), running, fast cycling, fast swimming, or playing sport (vigorous activity).The data are considered valid if the participants wear the Fitbit for ≥10 hours/day on ≥5 consecutive days (4 valid weekdays+1 valid weekend day). Higher minutes indicate more physically active.

SECONDARY OUTCOMES:
Healthy dietary intake | Change from baseline assessment to 12 weeks post-intervention
  The 8-item Starting-The-Conversation is a simplified food frequency instrument for identifying healthy and unhealthy dietary behaviours. Item scores are added to create a summary score (minimum score: 0; maximum score: 6), with higher summary scores reflecting the greatest room for improvement. The STC had acceptable construct validity and was found sensitive to change (Paxton et al., 2011)
Autonomous motivation | Change from baseline assessment to 12 weeks post-intervention
  The 19-item Chinese version of the Behavioural Regulation in Exercise Questionnaire-2 will be used to measure why the participants engage in physical activity by providing several possible reasons that represent varying degrees of motivation (19 items, 5-point Likert Scale). Item scores are added to create a summary score (minimum score: 0; maximum score: 76), with higher summary scores reflecting the greatest room for improvement. This instrument had adequate internal consistencies (α=.75), factorial validity and discriminant validity in Hong Kong university students (Chung et al. 2012).
Psychological flexibility | Change from baseline assessment to 12 weeks post-intervention
  The 7-item Chinese version of the Acceptance and Action Questionnaire-II. The scale of 1 (never true) to 7 (always true). Item scores are added to create a summary score (minimum score: 7; maximum score: 49), with higher summary scores indicating poor psychological flexibility (i.e., more psychologically inflexible) and a lower total score reflect high psychological flexibility. It demonstrated good internal consistencies (α = .88) and test-retest reliabilities (r = .79-.81) in adult populations in Hong Kong (Chong et al., 2019).
Mental status | Change from baseline assessment to 12 weeks post-intervention
  The 18-item Chinese version of the Brief Psychiatric Rating Scale will be used to assess the mental status of the participants. Items are rated on a 7-point Likert scale, from 1 = "not present" to 7 = "extremely severe". Items scores are added to create a summary score (minimum score: 18; maximum score: 126), with higher scores indicate poor mental health. This scale has been used globally in mental health services research, with previous studies indicating good content validity and internal consistency (α = .88) in people with mental illness in Hong Kong (Chien et al., 2015). A higher score suggests a greater level of psychopathology.
  .
Perceived quality of life | Change from baseline assessment to 12 weeks post-intervention
  The 26-item Chinese version of the World Health Organization Quality of Life-BREF will be adopted to assess the quality of life as perceived by patients, in terms of physical health, psychological health, social relationship and environmental quality of life. Responses to questions are on a 1-5 Likert scale where 1 represents "disagree" or "not at all" and 5 represents "completely agree" or "extremely". Items scores are added to create a summary score (minimum score: 26; maximum score: 130), with higher scores indicate stronger perceptions along with that question item. This instrument was modified from the World Health Organization Quality of Life-100, it has been shown to have satisfactory internal consistency and test-retest reliability among Chinese psychiatric patients (Leung et al., 1997).

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Yu CHONG, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, North District Hospital, Sheung Shui, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chong YY, Chien WT, Mou H, Ip CK, Bressington D. Acceptance and Commitment Therapy-based Lifestyle Counselling Program for people with early psychosis on physical activity: A pilot randomized controlled trial. Schizophr Res. 2025 Jan;275:1-13. doi: 10.1016/j.schres.2024.11.007. Epub 2024 Nov 28. PMID 39612765